CLINICAL TRIAL: NCT06594679
Title: A Study of Niraparib in Combination With Abemaciclib for Late Line Treatment of Ovarian Cancer: a Single Center, Open Label, Single Arm, Phase Ib/II Trial NICHOL TRIAL
Brief Title: A Study of Niraparib in Combination With Abemaciclib for Late Line Treatment of Ovarian Cancer (NICHOL TRIAL)
Acronym: NICHOL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: GlaxoSmithKline (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NICHOL INT 124/23
Record Dates: First submitted 2024-08-19; First posted 2024-09-19 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ARM 1 (Experimental): Niraparib+Abemaciclib
  Interventions: Drug: Niraparib Tosylate Monohydrate

INTERVENTIONS:
Drug: Niraparib Tosylate Monohydrate — Combination of niraparib and abemaciclib
  Other Names: Abemaciclib

SUMMARY:
This is an interventional trial. The goal of this clinical trial is dose finding. There are two phases: phase Ib to determine the MTD and recommended phase II dose of niraparib in combination with abemaciclib in patients with advanced ovarian cancer.

Target population will be patients (woman, age > 18 years) with epithelial ovarian, fallopian tube or peritoneal cancer treated with at least 2 lines of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Has read and understands the informed consent form and has given written informed consent prior to any study procedures.
* Age > 18 years
* Life expectancy of at least 3 months
* Histologically confirmed epithelial ovarian, primary peritoneal, or fallopian tube cancer
* Confirmed recurrent epithelial ovarian, primary peritoneal, or fallopian tube cancer for which there is no known or established treatment available with curative intent.
* Able to provide archived tumor tissue;(formalin fixed-paraffin embedded (FFPE) tumor sample or a minimum of 20 unstained slides is required for study eligibility.

NOTE: if archived tissue is not available, patient must be willing to undergo a tumor biopsy at screening if medically feasible.

* Patients must have completed at least 2 previous chemotherapy regimens for platinum sensitive disease (> 6 months). Patients must have completed their last therapy regimen > 4 weeks prior to treatment initiation and have radiological confirm of progression disease.
* Patients could have received maintenance therapy with a PARPi, but they must remain sensitive to platinum-based chemotherapy, based on the radiological or CA-125 response to their most recent course of platinum-based chemotherapy (carboplatin, cisplatin or oxaliplatin) or have demonstrated progressive disease while taking a PARP inhibitor as a previous therapy. Response to prior PARP inhibitor is not required.
* Prior PARP therapy could have been administered as either treatment for recurrent disease or as maintenance following prior treatment.
* Patients must have or agree to undergo tumor HRD testing and somatic BRCAmut status testing at screening.
* Patients must agree to undergo blood samples during screening and at the end of treatment for cytogenetic analysis.
* Phase 2 patients only: presence of measurable disease according to RECIST v1.1 criteria as assessed locally by Investigators.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-1.
* Absolute neutrophil count (ANC) ≥ 1500/L (within 14 days of study drugs initiation).
* Hemoglobin (Hgb) > 9 g/dL with no blood transfusion in the past 14 days (within 14 days of study drug[s] initiation).
* Platelets > 100,000/L (within 14 days of study drug[s] initiation) with no platelets transfusion in the past 14 days.
* Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 x upper limit of normal (ULN) or ≤ 5 x ULN if known hepatic metastases (within 14 days of study drugs initiation).
* Serum bilirubin within normal limits (WNL) or ≤ 1.5 x ULN in patients with liver metastases; or total bilirubin ≤ 2.0 x ULN with direct bilirubin WNL in patients with well documented Gilbert's syndrome (within 14 days of study drugs initiation).
* Patients should have calculated or measured creatinine clearance of ≥ 50 mL/min according to Cockroft-Gault.
* Willingness and ability to comply with study and follow-up procedures.
* Women of child-bearing potential must have a negative pregnancy test (serum) within 3 days prior to starting the study drug. Both males and females must agree to adequate birth control if conception is possible during the study and for 6 months after the last dose; in this case, patients must take a monthly pregnancy test for the duration of the study. Female patients are considered to not be of child-bearing potential if they have a history of tubal ligation or hysterectomy or are post-menopausal with a minimum of 1 year without menses.

The methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include:

* combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

  * oral;
  * intravaginal;
  * transdermal
* progestogen-only hormonal contraception associated with inhibition of ovulation:

  * oral;
  * injectable;
  * implantable.
* intrauterine device (IUD);
* intrauterine hormone-releasing system (IUS);
* bilateral tubal occlusion;
* vasectomised partner;
* sexual abstinence.

Additional inclusion criteria:

- Patients must agree to not donate blood during the study or for 90 days after the last dose of study treatment.

Exclusion Criteria:

* Any other prior therapy directed at the malignant tumor, including immunologic agents administered within 4 weeks prior to first dose of study drug
* Major surgical procedures ≤ 28 days of beginning study treatment, or minor surgical procedures < 7 days. No timeline window required for port-a-cath placement.
* Patients who received radiotherapy must have completed and fully recovered from the acute effects of radiotherapy. A washout period of at least 14 days is required between end of radiotherapy and randomization.
* History of any ≥ grade 3 hematological toxicity due to prior chemotherapy that persisted for more than 4 weeks.
* Patient has uncontrolled hypertension according to CTCAE v. 5.0
* Grade > 1 toxicity from prior therapy (except alopecia or anorexia) that contraindicates start of new treatment.
* Patient has inability to swallow oral medications or patients with gastrointestinal disorders likely to interfere with absorption of the study medication. Note: Patient may not have a percutaneous endoscopic gastrostomy (PEG) tube or be receiving total parenteral nutrition (TPN).
* Known central nervous system (CNS) disease other than neurologically stable, treated brain metastases - defined as metastasis having no evidence of progression or hemorrhage for at least 28 days after treatment (including brain radiotherapy). Must be off any systemic corticosteroids for the treatment of brain metastases for at least 14 days prior to enrollment.
* Chronic assumption of drugs or other products with a narrow therapeutic index and known to be CYP3A4 substrates, or drugs or other products known to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 2 weeks prior to day -3 of dosing and withheld throughout the study until 2 weeks after the last dose of study drug. Co-administration of aprepitant or fosaprepitant during this study is prohibited.
* Herbal preparations are not allowed throughout the study. These herbal medications include but are not limited to: St. John's wort, kava, ephedra (mahung), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto and ginseng, grapefruit and seville orange. Patients should stop using these herbal medications at least 7 days prior to first dose of study treatment.
* Any known hypersensitivity or contraindication to the components of the study drugs.
* Any of the following cardiac diseases currently or within the last 6 months: a. Unstable angina pectoris; b. Congestive heart failure; c. Acute myocardial infarction; d. Conduction abnormality not controlled with pacemaker or medication; e. Significant ventricular or supraventricular arrhythmias (patients with chronic rate- controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible).
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Evidence of corrected QT interval (specifically QTc calculated using the Fridericia formula [QTcF]) > 470 msec from a single electrocardiogram (ECG) performed at study entry or congenital or acquired long QT syndrome.
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea).
* Pregnant or breast-feeding. Female patients should not breastfeed or store milk within 30 days of receiving the final dose of niraparib and abemaciclib.
* Serious active infection at the time of study entry, or another serious underlying medical condition that would impair the ability of the patient to receive study treatment.
* Presence of other active invasive cancers (except for definitively treated in-situ carcinomas [e.g. breast, cervix, bladder, skin melanoma], or basal or squamous cell carcinoma of the skin) within the past 24 months.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with protocol.
* Patients with myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* History of human immunodeficiency virus (HIV) infection.
* History Active HBV or HCV infection. Patients whose disease is controlled under antiviral therapy are eligible. Testing for HBV or HCV is not necessary unless clinically indicated.
* History of cerebrovascular accident, PRES (posterior reversible encephalopathy syndrome), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* The patient has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, prior to randomization, or is currently enrolled in any other type of medical research (for example: medical device) judged by the sponsor not to be scientifically or medically compatible with this study.
* Pregnant or breast-feeding. Female patients should not breastfeed or store milk during the study treatment and within 30 days of receiving the final dose of niraparib and abemaciclib.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2027-09-18 (Estimated)

PRIMARY OUTCOMES:
dose finding | 18 months
  This is a dose-escalation study of niraparib plus abemaciclib followed by an efficacy study for late-line treatment of ovarian cancer
dose finding, phase Ib clinical trial | From enrollment to the end of phase 1
  Maximum tolerated dose (MTD) of niraparib in combination with abemaciclib in patients with advanced ovarian cancer defined as the dose level immediately below the dose at which ≥ 33% of patients experience dose-limiting toxicity as defined by protocol according to CTCAE 5.0
PART II: Disease control rate at 16 weeks (DCR16wks): | From enrollment of first patient of part II to to the 16-week-radiologic assessment of last patient
  proportion of patients whose disease shrinks (i.e. complete or partial response) or remains stable over 16 weeks after the start of niraparib + abemaciclib combination. Revised RECIST 1.1 criteria will be used to assess tumor response

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: No